CLINICAL TRIAL: NCT00610142
Title: Comparison of Atrophogenic Effect of Hydrocortison 1% Cream and Pimecrolimus 1% Cream Assessed by Optical Coherence Tomography (OCT) and 20-MHz Ultrasound of Uninvolved Skin in Patients With Atopic Dermatitis
Acronym: OCT-AD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TUD-OCT-AD-025
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; pimecrolimus; hydrocortison; Optical Coherence Tomography
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: pimecrolimus 1% cream
- 2 (Active Comparator)
  Interventions: Drug: hydrocortison 1% cream

INTERVENTIONS:
Drug: pimecrolimus 1% cream — twice a day one fingertip at a 2 times 2 cm2 area of uninvolved skin on the lateral forehead for 4 weeks
  Other Names: Elidel 1% cream
  Arms: 1
Drug: hydrocortison 1% cream — twice a day one fingertip at a 2 times 2 cm2 area of uninvolved skin on the lateral forehead for 4 weeks
  Other Names: Hydrogalen cream
  Arms: 2

SUMMARY:
to explore the atrophogenic potentials of hydrocortison 1% cream and pimecrolimus 1% cream on unaffected forehead skin

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years
* diagnosis of atopic dermatitis (Hanifin & Rajka Criteria)
* patients with atopic dermatitis not affecting the forehead

Exclusion Criteria:

* pregnancy / nursing mothers
* women in reproductive age without adequate contraception
* severe atopic dermatitis (IGA >= 4)
* UV-Therapy in past 4 weeks
* patients receiving any topical treatment on the face in past 6 month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
thickness of epidermis | 4 weeks

SECONDARY OUTCOMES:
thickness of dermis | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roland Aschoff, MD, Principal Investigator — Department of Dermatology, Medical Faculty, Technical University Dresden, Germany
Locations (1):
- Department of Dermatology, Medical Faculty, TU Dresden, Dresden, Germany

REFERENCES:
- [Result] Aschoff R, Schmitt J, Knuschke P, Koch E, Brautigam M, Meurer M. Evaluation of the atrophogenic potential of hydrocortisone 1% cream and pimecrolimus 1% cream in uninvolved forehead skin of patients with atopic dermatitis using optical coherence tomography. Exp Dermatol. 2011 Oct;20(10):832-6. doi: 10.1111/j.1600-0625.2011.01335.x. Epub 2011 Jul 19. PMID 21771098